CLINICAL TRIAL: NCT02432456
Title: Ketamine Infusion Therapy for the Management of Acute Pain in Adult Rib Fracture Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Nathan Kugler, Lead Research Resident, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO00024679
Record Dates: First submitted 2015-04-20; First posted 2015-05-04 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Wounds and Injuries; Rib Fractures
MeSH Terms: conditions — Wounds and Injuries; Rib Fractures | interventions — Ketamine; Acetaminophen; Ibuprofen; Pantoprazole; Methocarbamol; Analgesics, Opioid; Opiate Alkaloids; Narcotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Infusion (Placebo Comparator): Subjects in this arm will receive the institutional standard of care for rib fractures along with a placebo (NaCl) infusion.
  All patients will undergo Intercostal Nerve Blockade with administration of scheduled medications including acetaminophen, ibuprofen, pantoprazole, and methocarbamol. All subjects will receive adjunct opioids.
  Interventions: Drug: Placebo; Procedure: Intercostal Nerve Block; Drug: Acetaminophen; Drug: Ibuprofen; Drug: Pantoprazole; Drug: Methocarbamol; Drug: Opioid
- Ketamine Infusion (Experimental): Subjects in this arm will receive the institutional standard of care for rib fractures along with a ketamine infusion.
  All patients will undergo Intercostal Nerve Blockade with administration of scheduled medications including acetaminophen, ibuprofen, pantoprazole, and methocarbamol. All subjects will receive adjunct opioids.
  Interventions: Drug: Ketamine; Procedure: Intercostal Nerve Block; Drug: Acetaminophen; Drug: Ibuprofen; Drug: Pantoprazole; Drug: Methocarbamol; Drug: Opioid

INTERVENTIONS:
Drug: Ketamine — All individuals randomized to the experimental arm of the trial will receive early ketamine therapy (within 6 hours of admission) at a rate of 0.15 mg/kg/hr dosed based on ideal body weight. Individuals in the control arm will receive our standard of care for thoracic trauma patients, however, they will receive an additional placebo infusion of normal saline.
  Arms: Ketamine Infusion
Drug: Placebo — Individuals enrolled into the control arm of the trial will receive a normal saline placebo infusion at a rate equivalent to the dosage of ketamine in the experimental arm.
  Other Names: NaCl Placebo Solution
  Arms: Placebo Infusion
Procedure: Intercostal Nerve Block — All individuals enrolled into the trial will undergo an Intercostal Nerve Blockade as a part of the institutional standard of care for rib fractures. This procedure will be performed according to current standard protocols in the Emergency Department or on admission.
  Other Names: Rib Block
Drug: Acetaminophen — All patients admitted to the hospital will be placed on scheduled acetaminophen 1000mg PO q 6 hours unless signs of liver disease/impairment or creatinine clearance < 35ml/min at which point dosage would be reduced to 650mg q 8 hours. Individuals unable to take oral medications would be placed on intravenous acetaminophen.
  Other Names: Tylenol
Drug: Ibuprofen — All patients will be placed on scheduled Ibuprofen or an equivalent NSAID at dosage of 600mg every 6 hours. Patients must have a Glomerular Filtration Rate > 60 ml/min with no contraindications to NSAID therapy (e.g. Aspirin use, allergy/sensitivity, concurrent ACE inhibitor use, other nephrotoxins, etc)
  Other Names: Advil, Motrin
Drug: Pantoprazole — All individuals on scheduled Non-Steroidal Anti-Inflammatory Drug (NSAID) therapy will receive scheduled pantoprazole at 40mg daily. Individuals unable to take medications orally will be placed on intravenous therapy. Individuals with previous reaction or intolerance to pantoprazole will be placed on an equivalent proton pump inhibitor.
  Other Names: Protonix
Drug: Methocarbamol — All individuals enrolled in the trial will be placed on scheduled methocarbamol 500 mg orally every 6 hours while admitted. Individuals with previous intolerance to methocarbamol will be placed on a pharmacy directed equivalent.
  Other Names: Robaxin
Drug: Opioid — All individuals will receive as needed opiate therapy as an adjunct to the scheduled medications and "ketamine/placebo" solution. Choice in opiate therapy will be at the discretion of the attending trauma faculty. Dosage and adjustments will be in accordance with the institutional policy on appropriate opiate dosage adjustment.
  Other Names: opiate, narcotic

SUMMARY:
This study will evaluate the effectiveness of ketamine infusions in the management of acute pain resulting from broken ribs suffered following a blunt trauma. Half of patients will receive the institutional standard of care and a placebo infusion (no active medication). The other half of patients will receive the institutional standard of care and a ketamine infusion. All subjects and staff will be blinded as to whether they are receiving placebo or ketamine.

DETAILED DESCRIPTION:
A prospective randomized, double blinded trial of ketamine use in adult and elderly blunt trauma patients with associated rib fractures admitted to the trauma service will be conducted. Examples of blunt mechanisms include assault, falls, motor vehicle collisions, motorcycle crashes, motor vehicle pedestrian collisions, crush injuries, and bicycle accidents. The experimental arm of the trial will receive ketamine infusion therapy while the control arm receives saline placebo infusions at an equivalent rate. All patients will be managed with adjunct therapy including opiates in accordance with the institutional thoracic trauma protocols. Two separate trials based on patient age are included in this study. Elderly rib fracture patients are certainly of interest but will be evaluated as a distinct entity given the discrete differences in the complications of rib fractures and the goals of therapy.

All blunt trauma patients with associated rib fractures will be screened. All patients will be enrolled into the institutional standard thoracic trauma pathway. All individuals will undergo Intercostal Nerve Block (ICNB) in the Emergency Department or on admission to the Intensive Care Unit. In addition to scheduled medications per institutional thoracic trauma protocols, all patients will receive adjunct opiate therapy. Patients will be screened by the clinical and pharmacy staff following the diagnosis of rib fractures for eligibility. Patients enrolled into the trial will be randomized into either the experimental or control arm of the trial. The Investigational Drug Services (IDS) department will randomize all enrollees and handle administration of all trial drugs. The infusate will be mixed by the IDS department and all bags will be labeled "Ketamine / Placebo." The IDS department will have unique bag identifiers, which will allow them to identify which bags have active ketamine and which are placebo in case of emergency.

Patients will be randomized in a 1:1 fashion for experimental and control arms. Those enrolled in the experimental arm will receive early ketamine infusion therapy at a fixed infusion rate. For those enrolled in the adult trial the infusion rate will be 2.5 mcg/kg/min while those in the elderly trial will receive infusions at 2.0 mcg/kg/min. All ketamine infusions will be calculated based on ideal body weight (IBW), unless actual body weight is less than ideal. IBW will be calculated for males as 50kg + 2.3*(number of inches above 5 feet) and for women as 45.5kg + 2.3*(number of inches over 5 feet). Patients randomized to the control arm will receive placebo saline solution at an equivalent rate. Time zero will be defined as the time at which the "ketamine / placebo" infusion is begun. For inclusion in the trial, initiation of ketamine / placebo infusions must take place within 6 hours of presentation to Froedtert Memorial Lutheran Hospital (FMLH). Ketamine infusion therapy will be continued for 48 hours. At 6-8 hours post-ICNB all subjects will be assessed for need for repeat ICNB. Need for repeat ICNB will be defined by a thoracic specific numeric pain score greater than seven. Between eight and ten hours post-ketamine infusion initiation, subjects who have thoracic specific pain scores above seven will be evaluated for epidural placement by the Regional Anesthesia and Acute Pain Service.

A subject will be allowed to remove himself/herself from the trial or be un-blinded should he/she, pharmacy, anesthesia, and/or surgical staff deem it medically necessary. Medical necessity would be determined by inability to treat the patient appropriately without knowledge of trial assignment; otherwise the assumption of treating staff will be all patients have received ketamine. All adverse events will be recorded and if necessary subjects will be un-blinded in the event of a serious adverse event. The trauma and anesthesia teams along with the inpatient clinical pharmacists will monitor all trial patients for any adverse event trends. Patients will be followed through the time of discharge.

ELIGIBILITY:
Inclusion Criteria:

1. age greater than 18 years
2. rib fractures following recent trauma with admission to Froedtert Memorial Lutheran Hospital

Exclusion Criteria:

1. history of adverse reaction / intolerance to ketamine therapy
2. elevated intracranial pressure
3. ischemic heart disease defined as active acute coronary syndrome
4. severe, poorly controlled hypertension (Systolic Blood Pressure > 200 mmHg or Diastolic Blood Pressure > 100 mmHg)
5. current opiate agonist/antagonist therapy
6. concurrent use of monoamine oxidase inhibitors (MAOIs)
7. chronic pain or opioid tolerance defined as > 3 weeks of >30mg oral morphine equivalents per day
8. current substance abuse with opiates (prescription and/or heroin) or ketamine
9. Glasgow Coma Scale <13
10. Intubation on arrival or need for urgent intubation on arrival
11. inability to delineate pain and/or appropriately communicate with staff
12. history of psychosis
13. three or more psychotropic medications
14. active delirium
15. glaucoma
16. pregnancy
17. prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2015-09; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W Carver, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Carver TW, Kugler NW, Juul J, Peppard WJ, Drescher KM, Somberg LB, Szabo A, Yin Z, Paul JS. Ketamine infusion for pain control in adult patients with multiple rib fractures: Results of a randomized control trial. J Trauma Acute Care Surg. 2019 Feb;86(2):181-188. doi: 10.1097/TA.0000000000002103. PMID 30376537

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult Study: From August 2015 to December of 2017, all adult blunt trauma patients with three or more rib fractures were screened for eligibility in this study.
  Elderly Study: From August 2015 to June 2018, all elderly blunt trauma patients with three or more rib fractures were screened for eligibility in the study.
Pre-assignment Details: 153 patients agreed to participate. Three subjects (two from elderly and one from adult) were randomized but withdrawn prior to collecting any data or initiation of the infusions. This left a total of 150 participants within the trial, of which 75 were randomized to the placebo infusion with the other 75 randomized to the ketamine infusion.
Groups:
- Placebo Infusion: Subjects in this arm received the institutional standard of care for rib fractures along with a placebo (NaCl) infusion.
- Ketamine Infusion: Subjects in this arm will receive the institutional standard of care for rib fractures along with a ketamine infusion at a rate of 2.5 mcg/kg/min dosed based on ideal body weight.
Period: Overall Study
Arm/Group | Placebo Infusion | Ketamine Infusion
Started | 75 | 75
Completed | 75 | 75
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Infusion | Ketamine Infusion | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 45 | 91
  >=65 years | 29 | 30 | 59
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 26 | 47
  Male | 54 | 49 | 103
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 75 | 75 | 150
BMI [Median (Inter-Quartile Range); unit: kg/m^2] — Population: Adult trial consisted of 91 participants. The elderly trial consisted of 59 participants.
  kg/m^2
    Adult BMI: number analyzed (Participants) | 46 | 45 | 91
    Adult BMI | 28.5 [18.7 to 50] | 29 [18.3 to 51.7] | 29 [18.3 to 51.7]
    Elderly BMI: number analyzed (Participants) | 29 | 30 | 59
    Elderly BMI | 26.8 [20.6 to 39.7] | 29.2 [22.5 to 38] | 27.7 [20.6 to 39.7]
Number of Rib Fractures [Mean (Standard Deviation); unit: Rib Fractures] — Population: Adult trial consisted of 91 participants. The elderly trial consisted of 59 participants.
  Rib Fractures
    Adult: number analyzed (Participants) | 46 | 45 | 91
    Adult | 6.4 (3.3) | 6.4 (3.2) | 6.4 (3.2)
    Elderly: number analyzed (Participants) | 29 | 30 | 59
    Elderly | 6.5 (3.4) | 6.1 (2.6) | 6.3 (3.0)
Flail Chest [Number; unit: participants] — Population: Adult trial consisted of 91 participants. The elderly trial consisted of 59 participants.
  participants
    Adult: number analyzed (Participants) | 46 | 45 | 91
    Adult | 11 | 15 | 26
    Elderly: number analyzed (Participants) | 29 | 30 | 59
    Elderly | 9 | 4 | 13
Injury Severity Score, median [Median (Inter-Quartile Range); unit: Injury Severity Scale Score] — Population: Injury severity of each of 6 body systems is scored according the Abbreviated Injury Scale. Three body systems with the highest AIS scores are used to calculate the Injury Severity Score (ISS). These scores are squared and the results summed to produce the Injury Severity Score which ranges from 3-75. The higher the ISS the greater the injury.
  Injury Severity Scale Score
    Adult: number analyzed (Participants) | 46 | 45 | 91
    Adult | 13 [9 to 38] | 17 [9 to 34] | 14 [9 to 38]
    Elderly: number analyzed (Participants) | 29 | 30 | 59
    Elderly | 14 [9 to 48] | 13 [4 to 41] | 13 [4 to 48]
Injury Severity Score greater than15 [Number; unit: participants] — Population: Adult trial consisted of 91 participants. The elderly trial consisted of 59 participants.
  participants
    Adult: number analyzed (Participants) | 46 | 45 | 91
    Adult | 19 | 26 | 45
    Elderly: number analyzed (Participants) | 29 | 30 | 59
    Elderly | 14 | 10 | 24
ICU Admission [Number; unit: participants] — Population: Adult trial consisted of 91 participants. The elderly trial consisted of 59 participants.
  participants
    Adult: number analyzed (Participants) | 46 | 45 | 91
    Adult | 25 | 21 | 46
    Elderly: number analyzed (Participants) | 29 | 30 | 59
    Elderly | 26 | 25 | 51
Motor Vehicle Collision [Number; unit: participants] — Population: Adult trial consisted of 91 participants. The elderly trial consisted of 59 participants.
  participants
    Adult: number analyzed (Participants) | 46 | 45 | 91
    Adult | 20 | 21 | 41
    Elderly: number analyzed (Participants) | 29 | 30 | 59
    Elderly | 11 | 9 | 20
Fall [Number; unit: participants] — Population: Adult trial consisted of 91 participants. The elderly trial consisted of 59 participants.
  participants
    Adult: number analyzed (Participants) | 46 | 45 | 91
    Adult | 14 | 11 | 25
    Elderly: number analyzed (Participants) | 29 | 30 | 59
    Elderly | 14 | 16 | 30
Other Mechanism of Injury [Number; unit: participants] — Population: Adult trial consisted of 91 participants. The elderly trial consisted of 59 participants.
  participants
    Adult: number analyzed (Participants) | 46 | 45 | 91
    Adult | 12 | 13 | 25
    Elderly: number analyzed (Participants) | 29 | 30 | 59
    Elderly | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Numeric Pain Score
Description: Visual Analog Numeric Pain scores are reported as a single numeric score between 0 and 10. The more severe the pain the higher the number with 10 representing the most severe pain imaginable.
Time Frame: 12-24 hours post infusion
Population: Adult trial consisted of 91 participants. The elderly trial consisted of 59 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Infusion | Ketamine Infusion
Number analyzed (Participants) | 75 | 75
score on a scale
  Adult: number analyzed (Participants) | 46 | 45
  Adult | 6.1 (2) | 5.7 (2.1)
  Elderly: number analyzed (Participants) | 29 | 30
  Elderly | 5.2 (1.3) | 5.1 (1.9)

2. Secondary Outcome: Visual Analog Numeric Pain Score
Description: as for outcome 1
Time Frame: 24-48 hours post infusion
Population: Adult trial consisted of 91 participants. The elderly trial consisted of 59 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Infusion | Ketamine Infusion
Number analyzed (Participants) | 75 | 75
score on a scale
  Adult: number analyzed (Participants) | 46 | 45
  Adult | 5.8 (1.9) | 5.6 (2)
  Elderly: number analyzed (Participants) | 29 | 30
  Elderly | 4.4 (1.6) | 5.1 (1.7)

3. Secondary Outcome: Oral Morphine Equivalent (Narcotic Usage)
Description: This is an analysis of the narcotic utilization during the study. Oral Morphine Equivalents is a means of standardizing narcotic utilization given a multitude of different medications are utilized. Medications are standardized to units (milligrams) or oral morphine for a standardized comparison.
Time Frame: 12-24 hours post infusion
Population: Adult trial consisted of 91 participants. The elderly trial consisted of 59 participants.
Measure: Median (Full Range); unit: oral morphine equivalents
Arm/Group | Placebo Infusion | Ketamine Infusion
Number analyzed (Participants) | 75 | 75
oral morphine equivalents
  Adult: number analyzed (Participants) | 46 | 45
  Adult | 45.0 [0 to 295] | 45 [0 to 187.2]
  Elderly: number analyzed (Participants) | 29 | 30
  Elderly | 30 [0 to 131] | 21.3 [0 to 203]

4. Secondary Outcome: Oral Morphine Equivalent (Narcotic Usage)
Description: as for outcome 3
Time Frame: 24-48 hours post infusion
Population: Adult trial consisted of 91 participants. The elderly trial consisted of 59 participants.
Measure: Median (Full Range); unit: oral morphine equivalents
Arm/Group | Placebo Infusion | Ketamine Infusion
Number analyzed (Participants) | 75 | 75
oral morphine equivalents
  Adult: number analyzed (Participants) | 46 | 45
  Adult | 67 [0 to 1201.0] | 69.0 [0 to 656.5]
  Elderly: number analyzed (Participants) | 29 | 30
  Elderly | 44 [0 to 302] | 25 [0 to 765]

5. Secondary Outcome: Length of Stay
Description: Total hospital length of stay in days up to 365 days.
Time Frame: Total Index Hospitalization up to 365 days
Population: Adult trial consisted of 91 participants. The elderly trial consisted of 59 participants.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo Infusion | Ketamine Infusion
Number analyzed (Participants) | 75 | 75
days
  Adult: number analyzed (Participants) | 46 | 45
  Adult | 4.0 [1 to 33] | 5 [1 to 20]
  Elderly: number analyzed (Participants) | 29 | 30
  Elderly | 6 [2 to 109] | 5 [2 to 50]

6. Secondary Outcome: Regional Anesthesia Utilization
Description: This is a measure of the Epidural Placement rates. Epidural placement was binary as in patient received or did not receive an epidural infusion catheter for supplemental pain management.
Time Frame: Total Index Hospitalization up to 365 days
Population: Adult trial consisted of 91 participants. The elderly trial consisted of 59 participants.
Measure: Number; unit: participants
Arm/Group | Placebo Infusion | Ketamine Infusion
Number analyzed (Participants) | 75 | 75
participants
  Adult: number analyzed (Participants) | 46 | 45
  Adult | 3 | 7
  Elderly: number analyzed (Participants) | 29 | 30
  Elderly | 6 | 4

7. Secondary Outcome: Respiratory Failure
Description: Respiratory failure within this trial was defined by the need for unanticipated intubation and/or transfer to ICU for respiratory support.
Time Frame: Total Index Hospitalization up to 365 days
Population: Adult trial consisted of 91 participants. The elderly trial consisted of 59 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Infusion | Ketamine Infusion
Number analyzed (Participants) | 75 | 75
Participants
  Adult: number analyzed (Participants) | 46 | 45
  Adult | 3 | 2
  Elderly: number analyzed (Participants) | 29 | 31
  Elderly | 0 | 0

8. Secondary Outcome: Hallucination
Description: Hallucinations were documented and confirmed by the treating medical team.
Time Frame: Total Index Hospitalization up to 365 days
Population: Adult trial consisted of 91 participants. The elderly trial consisted of 59 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Infusion | Ketamine Infusion
Number analyzed (Participants) | 75 | 75
Participants
  Adult: number analyzed (Participants) | 46 | 45
  Adult | 1 | 0
  Elderly: number analyzed (Participants) | 29 | 30
  Elderly | 2 | 2

9. Secondary Outcome: Oral Morphine Equivalent (Narcotic Usage) in Severely Injured
Description: as for outcome 3
Time Frame: Total Index Hospitalization up to 365 days
Population: A total of 45 participants were categorized as severely injured within the adult trial. A total of 24 participants were categorized as severely injured within the elderly trial.
Measure: Median (Full Range); unit: oral morphine equivalents
Arm/Group | Placebo Infusion | Ketamine Infusion
Number analyzed (Participants) | 33 | 36
oral morphine equivalents
  Adult: number analyzed (Participants) | 19 | 26
  Adult | 170.5 [0 to 1589.0] | 153.0 [0 to 758.5]
  Elderly: number analyzed (Participants) | 14 | 10
  Elderly | 86.8 [0 to 376] | 67.5 [0 to 988]

ADVERSE EVENTS:
Time Frame: Data was collected for the duration of all participants hospitalizations. At time of discharge adverse event recording was stopped as patients were monitored throughout only their index stay defined up to 365 days.
Description: All adverse events were reported and reviewed by the IRB at our insitution.
Arm/Group | Placebo Infusion | Ketamine Infusion
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/75
Other Adverse Events (participants affected / at risk) | 15/75 | 7/75
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Infusion (N=75) | Ketamine Infusion (N=75)
Delirium (Psychiatric disorders) | 3 | 1 — Delirium as outlined by positive CAM testing
Sedation (Psychiatric disorders) | 6 | 2 — Concern on nursing that patient was sedated as result of over medication
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 | 2 — Need for intubation
Hallucinations (Psychiatric disorders) | 3 | 2

LIMITATIONS AND CAVEATS:
NPS presents challenges as pain is subjective and difficult to assess. Treating providers were allowed any medications within the multimodal rib fracture pain protocol leading to non-standardized pain regimens based on providers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT02432456/Prot_SAP_000.pdf